CLINICAL TRIAL: NCT01377337
Title: Does the Early Use of Sodium Bicarbonate Improve Results of Cardiopulmonary Resuscitation Following Out-of-Hospital Cardiac Arrest - a Prospective, Controlled Clinical Trial
Brief Title: Sodium Bicarbonate in Cardiopulmonary Resuscitation
Acronym: SB CAT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0013-09-RMB
Record Dates: First submitted 2011-06-16; First posted 2011-06-21 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Sudden Cardiac Arrest
Keywords: cardiac arrest; cardiopulmonary resuscitation; (sodium) bicarbonate; return of spontaneous circulation; outcome
MeSH Terms: conditions — Death, Sudden, Cardiac; Heart Arrest | interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium bicarbonate (Active Comparator): 1 mEq/kg sodium bicarbonate administered intravenously immediately following the administration of the first epinephrine dose during advanced CPR.
  Interventions: Drug: sodium bicarbonate
- 0.9% NaCl (Placebo Comparator): 1 ml/kg of 0.9% NaCl (Blinded label)
  Interventions: Drug: sodium bicarbonate

INTERVENTIONS:
Drug: sodium bicarbonate — 1 mEq/kg sodium bicarbonate administered intravenously immediately following the administration of the first epinephrine dose during advanced CPR. Dose may be repeated every 5-10 minutes up to 3 doses.
  Note: The Placebo Arm receives 1 ml/Kg of 0.9% NaCl (in a blinded fashion).

SUMMARY:
Out-of-hospital cardiac arrests (OHCA) account for over 60% of deaths from coronary artery disease. The annual incidence of OHCA treated by Emergency Medical Systems (EMS) is 41-89 per 100,000 population. Outcome of OHCA and cardiopulmonary resuscitation (CPR) is very poor: Less than 1/3 of the victims regain spontaneous circulation (ROSC), 40-60% of those achieving ROSC suffer significant neurological disability due to brain hypoxia and only 1.7-6.4% are discharged from the hospital. In order to minimize hypoxia time, the primary goal of CPR is to achieve return of spontaneous circulation (ROSC) as fast as possible. Metabolic (lactic) acidosis develops rapidly during CA and is considered detrimental to CPR outcome. Sodium bicarbonate (SB), a generic, commonly used acid buffer, was subjected only to a single, small, prospective controlled trial that found a trend towards improved outcome in prolonged OHCA and CPR. Another study indicated that EMS's that used SB early and often during CPR had significantly higher ROSC rates and better long-term outcome compared with EMS's that used SB more seldom and administered it late in the course of CPR.

Aim of the Study:

To determine whether early administration of SB during OHCA and CPR improves short-term CPR outcome.

DETAILED DESCRIPTION:
General: Prospective, randomized, double blinded, placebo-controlled clinical trial. Exception from Informed Consent, under the regulations for the conduction of research in emergency situations, has been approved by the Helsinki Committee of the Rambam Medical Center and by the Supreme Helsinki Committee of the Israeli Ministry of Health. Included will be adult patients who suffer an OHCA, who do not respond to basic CPR and to early defibrillation and in whom advanced CPR is initiated. 1st dose (1 mEq/Kg) of SB/placebo will be administered by Israeli Magen David Adom (MDA) advanced life support (ALS) teams immediately following the first IV epinephrine. SB/placebo vials or syringes will be masked and coded. Calculated sample size is 2130 patients. Study endpoints include only short-term outcome variables - rates of ROSC and of admission to the emergency room.

Expected results: Based on previous analysis we expect a 20% improved short-term outcome in the SB treated group. Sample size was calculated accordingly.

Importance: Around 2.2 million OHCA's are treated by EMS worldwide annually. Current ROSC rate is ca. 30%. A 20% better short-term outcome will result in over 130,000 additional patients regaining spontaneous circulation annually.

Probable implications to Medicine: The use of SB in CPR is controversial. Current International Guidelines for CPR present very reserved recommendations regarding SB use. Results of this study may have a direct impact on the Guidelines and on the conduction of CPR world-wide. Based on the results of this trial, a Phase II trial, researching the effects of early SB administration on long-term outcome (hospital discharge and final neurological outcome) may be warranted and conducted.

ELIGIBILITY:
Inclusion Criteria:

* patients who suffer Out of hospital, non-traumatic cardiac arrest
* patients who do not respond to the initial resuscitation efforts (including basic CPR, defibrillation (when indicated) and other appropriate ACLS measures)
* patients in whom a vascular access (either an IV line or an intraosseous needle) has been obtained
* patients who have reached the "drugs" step in the ACLS algorithm.

Exclusion Criteria:

* Patients with known terminal illness
* Patients with a Do Not Resuscitate (or similar) order
* Cardiac arrest due to trauma, drug overdose or known intracranial disease
* Age less than 18 years
* Known pregnancy
* Patients in whom 30 minutes or more have passed from collapse to initiation of CPR
* If collapse time is unknown - patients with obvious death marks
* Patients with no vascular access (either an IV line or an intraosseous needle)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2130 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Short-term survival | at completion of CPR
  proportion of patients who achieve return of spontaneous circulation (ROSC) and proportion of patients admitted alive (not requiring CPR) to the hospital's emergency room

CONTACTS AND LOCATIONS:
Overall Officials: Gad Bar-Joseph, Principal Investigator — Rambam Health Care Campus
Locations (2):
- Israel (2):
  - Rambam Medical Center, Haifa
  - Magen David Adom, Tel Aviv